CLINICAL TRIAL: NCT03655197
Title: Lipidome and Microbiome Profile of the Eye in Rosacea
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1138313
Record Dates: First submitted 2018-08-21; First posted 2018-08-31 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Rosacea; Ocular Rosacea; Cutaneous Rosacea
Keywords: Microbiome; Lipidome
MeSH Terms: conditions — Rosacea | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: Healthy Subjects-No Intervention Ocular Rosacea Subjects-Mandatory Doxycycline Intervention Cutaneous Rosacea Subjects-Optional Doxycycline Intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Subjects (No Intervention): Healthy subjects will receive no intervention and will have samples collected only at one visit after Dove soap washout.
- Ocular Rosacea Subjects (Experimental): Ocular rosacea subjects will receive mandatory Doxycycline intervention and will have samples collected at two visits, before starting intervention and at the completion of the intervention.
  Interventions: Drug: Doxycycline
- Cutaneous Rosacea Subjects (Other): Doxycycline intervention is optional for cutaneous rosacea subjects. If they do not participate, samples will only be collected at one visit after Dove soap washout. If they do decide to participate, samples will also be collected after completion of the Doxycycline intervention.
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — For those participating in the Doxycycline intervention, they will take 100 mg twice daily for 1 month.
  Arms: Cutaneous Rosacea Subjects; Ocular Rosacea Subjects

SUMMARY:
The question that the investigators aim to address in this proposal is how the local lipid mediator profiles of ceramides and eicosanoids are altered in cutaneous and ocular rosacea and how antibiotics alter the lipidome. The investigators also seek to understand how the microbiome is changed in those with and without rosacea, and how the microbiome is altered in those with rosacea. Understanding how the lipidome is modulated in rosacea with antibiotic treatment will serve as the first step in targeting therapies toward directly altering the lipidome to reduce inflammation and ultimately reduce the use of antibiotics.

DETAILED DESCRIPTION:
Rosacea is a common condition that has multiple subtypes that exhibit inflammation and deficits in the skin/eye barrier function. Cutaneous rosacea is estimated to have an incidence of 10-22% while the prevalence of ocular rosacea ranging from 6-72%. Although rosacea is not an infection, antibiotics are widely used as first-line therapy due to their anti-inflammatory and skin-barrier function supporting effects. The most common class of antibiotics used are the tetracyclines, such as doxycycline and minocycline. With the emergence of community acquired methicillin resistant Staphylococcus aureus (MRSA) as well as macrolide resistant Streptococci and Staphylococci, there is growing concern for the widespread use of antibiotics for non-infectious conditions.

The current clinical gap in practice is that there are few alternative therapies to antibiotics and this is partly due to our lack of understanding of what leads to the impaired skin/eye barrier and inflammation in rosacea. Few lipid-based studies have been performed in rosacea but there is early evidence for the importance in the lipidome to rosacea. The sebum in those with papulopustular rosacea was identified to have an abnormal profile to their sebum with a deficiency in long chain saturated fatty acids6 that correlates with the deficient skin barrier that is seen in rosacea. Treatment with minocycline was shown to restore skin barrier function in papulopustular rosacea but no lipid profile related measures were performed. Moreover, no studies have evaluated the role of other lipid mediators that are closely associated with the skin barrier and inflammation such as the ceramides and the eicosanoids.

The question that the investigators aim to address in this proposal is how the local lipid mediator profiles of ceramides and eicosanoids are altered in cutaneous and ocular rosacea and how antibiotics alter the lipidome. The investigators also seek to understand how the microbiome is changed in those with and without rosacea, and how the microbiome is altered in those with rosacea. Understanding how the lipidome is modulated in rosacea with antibiotic treatment will serve as the first step in targeting therapies toward directly altering the lipidome to reduce inflammation and ultimately reduce the use of antibiotics.

ELIGIBILITY:
Inclusion Criteria for subjects:

* Aged 18 and older
* Subjects that meet one of the following criteria:

  * Healthy subjects without an inflammatory facial rash or an inflammatory eye condition
  * Subjects diagnosed with ocular rosacea or cutaneous rosacea (papulopustular or erythematotelangiectatic) by either a board-certified dermatologist or ophthalmologist

Exclusion Criteria

* Those who are prisoners or cognitively impaired.
* Those who have had any change to their hormonal birth control regimen in the last 4 weeks
* Systemic antibiotic use in the last four weeks
* Allergy or known intolerance to tetracyclines
* Those who wear contact lenses
* Autoimmune disease such as lupus, dermatomyositis that has cutaneous involvement
* Those who are pregnant or may become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Lipidome Change in Diversity | 1-5 weeks
  Lipid profiles will be assessed, such as inflammatory and non-inflammatory lipid mediators, along with the alpha and beta diversity of the lipidome of the samples. The shifts in diversity of the lipidome will be quantified.
Microbiome Change in Diversity | 1-5 weeks
  The microbiome content and the microbiome between sites on the same patient will be assessed. The assessment will examine what new bacteria becomes present.
Lipidome Change in Quantity | 1-5 weeks
  Lipid profiles will be assessed, such as inflammatory and non-inflammatory lipid mediators, along with the alpha and beta diversity of the lipidome of the samples. The increase or decrease of inflammatory and non-inflammatory lipid mediators will be quantified.
Microbiome Change in Quantity | 1-5 weeks
  The microbiome content and the microbiome between sites on the same patient will be assessed. The assessment will examine how the previously present bacteria changes in quantity.

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD, MS, Principal Investigator — UC Davis, Department of Dermatology; Mark Mannis, MD, Principal Investigator — UC Davis, Department of Ophthalmology
Locations (1):
- University of California-Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No